CLINICAL TRIAL: NCT05401513
Title: Effects of an Exercise Program Based on the Pilates Method in Brazilian Air Force Helicopter Pilots With Low Back Pain: Randomized Controlled Trial
Brief Title: Pilates Method in Helicopter Pilots With Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Jamilson Simões Brasileiro, Professor, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LCCB2022
Record Dates: First submitted 2022-05-29; First posted 2022-06-02 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Low Back Pain
Keywords: low back pain; physiotherapy; muscle fatigue
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates Group (Experimental): 12-weeks exercise program, twice a week, with Pilates method exercises.
  Interventions: Other: Pilates Group
- Control Group (No Intervention): 12-weeks maintaining their normal physical activity routine.

INTERVENTIONS:
Other: Pilates Group — The individuals of the Pilates group will perform specific exercises of the method, which will involve mobility, stability and muscular resistance. The exercises will progress according to the level of difficulty (basic, intermediate and advanced), load and repetition every three or four weeks.
  Arms: Pilates Group

SUMMARY:
The purpose of this study is to analyze the effects of an exercise program, based on the Pilates method, on the low back pain and muscle fatigue of Brazilian Air Force helicopter pilots.

DETAILED DESCRIPTION:
Methods: This is a randomized controlled trial composed by Brazilian Air Force helicopter instructors. The volunteers will be submitted to an initial evaluation composed by painful sensation, analyzed through the Numerical Pain Scale, disability associated with low back pain, using the Roland Morris Disability Questionnaire, and back muscle fatigue, through the Ito test. The pilots will be randomly assigned to the Exercise Group (exercise program based on the Pilates method, twice a week for 12 weeks) and Control Group (no intervention). After the sixth and 12th week of the beginning of the intervention program a new evaluation will be carried out, identical to the initial one.

ELIGIBILITY:
Inclusion Criteria:

* Brazilian Air Force helicopter instructors - Natal Air Base;
* Nonspecific low back pain for more than 3 months with a score of 2 or more at Numerical Pain Rating Scale.

Exclusion Criteria:

* Be undergoing physiotherapeutic treatment during the study period;
* Corticosteroids treatment in the last two weeks;
* Anti-inflammatory treatment in the previous 72 hours;
* Have specific spinal pathologies, such as spondylitis, spondylolysis, spondylolisthesis, disc herniation with radiculopathy or those who have had spinal surgery in the last year or who have a recent history of spinal fracture.

Ages: 20 Years to 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-06-20 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Painful sensation | Change from baseline in low back pain sensation at 6 weeks and 12 weeks after the intervention protocol
  To compare the painful sensation in the lumbar region using the Numerical Pain Rating Scale (NPRS) across a range of 11, with 0 being described as 'no pain' and 10 as 'worst possible pain'.

SECONDARY OUTCOMES:
Functional disability associated to back pain | Change from baseline in disability at 6 weeks and 12 weeks after the intervention protocol
  To analyze the self-report low back pain disability through the Roland Morris Disability questionnaire.
Back muscle fatigue | Change from baseline in back muscle fatigue at 6 weeks and 12 weeks after the intervention protocol
  Measure the back muscular resistance to fatigue using the Ito test

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Rio Grande do Norte, Natal, Rio Grande do Norte, Brazil